CLINICAL TRIAL: NCT05714995
Title: Evaluation of the Therapeutic Approach of Aromatherapy by Olfaction of Essential Oils in Association With Hypnosis in the Care of Patients Followed in Oncology for Cancer Within a Mobile Palliative Care Support Team (EMASP)
Brief Title: Evaluation of the Therapeutic Approach of Aromatherapy by Olfaction of Essential Oils in Association With Hypnosis in the Management of Patients Followed for Cancer
Acronym: HYPNO-AROMA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: HYPNO-AROMA
Record Dates: First submitted 2023-01-12; First posted 2023-02-06 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Hypnosis; Aromatherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypnosis: patients in the hypnosis group will perform self-hypnosis sessions
  Interventions: Other: hypnosis
- hypnosis with aromatherapy: patients in the hypnosis with aromatherapy group will perform self-hypnosis sessions with inhalation of an essential oil
  Interventions: Other: Hypnosis with aromatherapy

INTERVENTIONS:
Other: hypnosis — The hypnosis session involves the following steps:
  1. Preparation for the activation of the hypnotic trance
  2. Activation of the hypnotic trance
  3. Deepening the hypnotic trance
  4. Maintaining hypnotic trance
  5. Coming out of the hypnotic trance
  Groups: hypnosis
Other: Hypnosis with aromatherapy — for patients in the hypnosis with aromatherapy group, before starting the hypnosis session, they will first choose an essential oil among the 5 proposed.
  They will pour a drop on their wrist then they will rub it and inhale deeply.
  The hypnosis session involves the following steps:
  1. Preparation for the activation of the hypnotic trance
  2. Activation of the hypnotic trance
  3. Deepening the hypnotic trance
  4. Maintaining hypnotic trance
  5. Coming out of the hypnotic trance
  Groups: hypnosis with aromatherapy

SUMMARY:
Patients having the following gestures (blood test, change of dressing for cancerous lesion and complete toilet in bed) will be identified by the team of the medical oncology department.

During the first contact (V0), the study will be presented to the patients in order to obtain their consent. Anxiety and well-being will be assessed before performing the gesture causing discomfort (gesture No.1). The gesture will then be performed and the patient's comfort will be evaluated after the gesture is performed in order to obtain the starting data for the study.

Patients will be reviewed in consultation according to the time recommended for each type of gesture.

During the second contact V1 (between 1 and 9 days after D0) anxiety and well-being will be assessed before performing the gesture causing discomfort (gesture No.2). Patients will then be randomized. After randomization, the first hypnosis session will be performed at the same time as gesture No. 2 and the patient's comfort will be evaluated after the gesture is performed. The patient will receive the self-hypnosis training on the same day.

A period of 7 ± 2 days will be considered for the learning time of self-hypnosis.

The third contact will take place on day D7+/-2 after V1. During this visit, anxiety and well-being will be assessed before performing the gesture causing discomfort (gesture No.3). Gesture No.3 will be carried out under the effect of self-hypnosis ± aromatherapy and the measurement of comfort will be carried out immediately afterwards

DETAILED DESCRIPTION:
Include (V0):

Patients in whom the following procedures must be performed:

* Blood samples via a central catheter with a percutaneous implantable chamber, with a Huber needle
* Peripheral venous samples
* Tumor Lesion Dressing
* Complete toilet in bed will be identified by the team of the medical oncology department. During the first contact (V0), the study will be presented to the patients in order to obtain their consent. After signing the consent and before performing the gesture causing discomfort (gesture No.1), anxiety and well-being will be assessed by the verbal administration of the ESAS scale. The gesture will then be performed and the patient's comfort will be assessed using the ESAS scale after the gesture has been performed in order to obtain the data at the start of the study. An appointment for the V1 visit (between 1 and 9 days after D0) will be set for the next procedure.

First V1 hypnosis session (between 1 and 9 days after D0):

During the second contact at visit V1 (between 1 and 9 days after D0), anxiety and well-being will be assessed before performing the gesture causing discomfort (gesture No.2). Randomization will take place immediately before performing the procedure. After randomization, the first session of hypnosis +/- aromatherapy will be performed at the same time as gesture No. 2 and the patient's comfort will be evaluated after the gesture is performed. During this hypnosis session, the patient will receive self-hypnosis training according to the group they belong to (self-hypnosis vs self-hypnosis + aromatherapy). An appointment for the realization of the next gesture (gesture No.3) will be set for D7 (+/- 2 days after V1). This period of time (7±2 days) will be considered the learning time for self-hypnosis.

Second V2 hypnosis session (D7+-/ 2 days after V1):

The third contact V2 will take place at (D7+/- 2 days after V1). During this visit, anxiety and well-being will be assessed before performing the gesture causing discomfort (gesture No.3). Gesture No.3 will be carried out under the effect of self-hypnosis ± aromatherapy and the measurement of comfort will be carried out immediately afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Patients followed in medical oncology and by the mobile palliative care support team
* From the first line of chemotherapy
* Patient requiring one of the following procedures:
* Blood samples via a central catheter with a percutaneous implantable chamber, with a Huber needle
* Peripheral venous samples
* Change of dressing for cancerous lesion
* Complete toilet in bed
* Patients who have given their consent
* Patient affiliated with a social security scheme

Exclusion Criteria:

* Protected person under guardianship or curatorship,
* Person deprived of liberty
* Person unable to express consent
* Pregnant woman and breastfeeding woman
* History of allergy or intolerance to essential oils
* Patients with cognitive or language disorders that make it impossible to answer the questionnaires
* Psychotic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients coming to HDJ or hospitalized in a conventional medical oncology unit, monitored from the 1st line of chemotherapy and taken care of by the mobile palliative care support team (EMASP)
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
difference in comfort score between the two groups: The comfort score will be evaluated by the French version of the pain scale of the Edmonton Symptom Assessment System | betwen the baseline and day 17
  The comfort score will be evaluated by the French version of the pain scale of the Edmonton Symptom Assessment System. The severity of each symptom was rated from 0 to 10 (0 = no symptom, 10 = worst possible intensity

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal de Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No